CLINICAL TRIAL: NCT03025841
Title: Population Pharmacokinetic (PK) Study of Zinforo (Ceftaroline) in Critical Care Patients With Early-onset Pneumonia and Normal or Augmented Renal Clearance
Acronym: CEFTAREA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEFTAREA
Record Dates: First submitted 2016-12-06; First posted 2017-01-20 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Ceftaroline

ARMS (1):
- Ceftaroline (Other): Patients receive Ceftaroline 600mg BID
  Interventions: Drug: Ceftaroline

INTERVENTIONS:
Drug: Ceftaroline

SUMMARY:
Pneumonia is the most frequent infection in critically ill patients and remains a significant challenge to intensivists world-wide due to persisting high mortality and morbidity. Compelling evidence suggests that appropriate antibiotic therapy remains the most important intervention to improve patients' outcome, including the administration of a suitable molecule at an optimized dosage regimen. A vast array of pathophysiological changes can occur in critically ill patients that can complicate antibiotic dosing. Knowledge of the pharmacokinetic and pharmacodynamic properties of the antibiotics used for the management of critically ill patients is essential for selecting the antibiotic dosing regimens, which will optimize patient outcomes. Changes in volume of distribution (Vd) and clearance (CL) of antibiotics have been noted in these patients, which may affect the antibiotic concentration at the target site. It follows that the pharmacodynamic parameters that determine antibiotic efficacy, which can vary between antibiotic classes, may also be affected. Optimization of these parameters is necessary to maximize the rate of response through patient recovery and minimized antibiotic resistance.

In a multicenter observational study in critically ill patients with normal plasma renal indices at admission, about 65% of patients manifested augmented creatinine clearance on at least one occasion in the first seven study days. Augmented creatinine clearance may significantly impact drug pharmacokinetics for a variety of renally eliminated pharmaceuticals (such as low-molecular weight heparins, aminoglycosides, glycopeptides, and β-lactams), leading to subtherapeutic concentrations and potentially adverse clinical outcomes. Currently little data exist that describe the consequences of augmented creatinine clearance on antibiotics PK.

Ceftaroline (600 mg bid) is a cephalosporin with expanded gram-positive activity, including MRSA and penicillin-resistant streptococcus, which was approved by the US Food and Drug Administration (FDA) on October 29, 2010 for the treatment of acute bacterial SSSIs and community-acquired bacterial pneumonia. Ceftaroline showed also good activity against some of the common gram-negative respiratory pathogens (eg, Haemophilus influenzae, Moraxella catarrhalis, Neisseria meningitidis, and Pasteurella multocida). However, it does not display clinically relevant activity against Pseudomonas aeruginosa, Stenotrophomonas maltophilia, or Acinetobacter baumannii. Ceftaroline also lacks activity against gram-negative organisms with extended-spectrum β-lactamases. Importantly, because ceftaroline appears to induce AmpC β-lactamases despite MIC values in susceptible range, ittheoretically should be avoided in gram-negative bacteria known to harbor inducible AmpC β-lactamases (eg, Serratia, Proteus, Citrobacter, Morganella, Enterobacter, Providencia, and P. aeruginosa). In patients, ceftaroline is given as a prodrug, ceftaroline fosamil. After intravenous administration, the prodrug is rapidly transformed by plasma phosphatase enzymes to its bioactive metabolite. The pharmacokinetics of ceftaroline has been evaluated in single and multiple dose studies in healthy volunteers, in subjects with various degrees of renal impairment and in healthy elderly subjects. The volume of distribution is equal to 20.3 L, which corresponds to extracellular fluid volume. The protein binding is low (20%). The main route of elimination is via renal excretion, with a clearance estimated to160 mL/min close to the creatinine clearance. The elimination half-live is 2.6 h in adults with normal renal function. Unfortunately, no PK study has been performed in infected critically ill patients with augmented creatinine clearance. The best PK-PD index predicting drug efficacy is %Time>CMI. A bacteriostatic effect is achieved when free drug concentrations exceed the MIC for 30 to 40% of the dose administration interval (30 to 40%T>MIC). Near maximum organism kill is achieved at 50 to 60%T>MIC (30%T>MIC for Staphylococcus aureus).

This project aims to characterize ceftaroline PK in patients with early-onset pneumonia and augmented creatinine clearance. The choice of ceftaroline is justified by its spectrum suitable for micro-organisms commonly encountered in early onset pneumonia, including methicillin-resistant Staphylococcus aureus. Secondary main objective is to predict the probably of reaching PK-PD targets using Monte Carlo simulations under various scenario in order to identify optimal ceftaroline administration schemes in critical care patients with various degrees of renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in ICU
* Under mechanical ventilation
* Developing early-onset (during the seven days following hospital admission) pneumonia caused by Gram positive and/or Gram negative bacteria.
* Having an augmented or normal renal clearance defined by a directly measured creatinine clearance, using MD-RD:

  * normal clearance: between 80 and 130 mL/min/1.73m²
  * augmented clearance: more than or equal to 130 mL/min/1.73m²

Exclusion Criteria:

* Having one or more risk factors of multi drug resistant bacteria:

  * antibiotic treatment in last 3 months
  * high level resistance in the unit
  * immunosuppression
  * one or more pneumonia risks factors, whose one hospitalization of more than 48 hours in past 90 days,
  * living in medical care house,
  * chronic hemodialysis,
  * home based wound care
  * resistant bacteria in the family environment
* Morbidly obese subjects (BMI>40 kg/m²)
* Septic shock
* Ceftaroline administered in past 14 days before inclusion
* Diuretic treatment
* Suspicion or confirmation pneumonia ceftaroline-resistant bacteria
* Known hypersensitivity due to Ceftaroline or cephalosporin antibiotics
* Known hypersensitivity due to Gentamicin or aminoglycosides antibiotics
* Hypersensitivity due beta lactamin antibiotics
* Anemia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Minimum plasma concentration of Ceftaroline | Day 6
Maximum plasma concentration of Ceftaroline | Day 6
Volume of distribution of Ceftaroline in plasma | Day 6
Clearance of Ceftaroline in plasma | Day 6
Elimination half life of Ceftaroline in plasma | Day 6

SECONDARY OUTCOMES:
Pharmacokinetic measures outcomes to obtain the dosing regimens through the monte carlo simulation. | Day 6
  in at least 90% of simulated subjects for minimal inhibitory concentration from 0.008 to 32 mg/L
Clinical efficacy during Ceftaroline treatment and two weeks after end of it | Day 28
  Patients will be considered to have clinical failure if they will have no response to the study drug on the basis of ongoing signs and symptoms of infection. Otherwise, patients will be considered to have clinical success
Safety evaluation by adverse events and serious adverse events collection | One month following the last administration

CONTACTS AND LOCATIONS:
Locations (1):
- CHU poitiers, Poitiers, France

REFERENCES:
- [Derived] Chauzy A, Gregoire N, Ferrandiere M, Lasocki S, Ashenoune K, Seguin P, Boisson M, Couet W, Marchand S, Mimoz O, Dahyot-Fizelier C. Population pharmacokinetic/pharmacodynamic study suggests continuous infusion of ceftaroline daily dose in ventilated critical care patients with early-onset pneumonia and augmented renal clearance. J Antimicrob Chemother. 2022 Oct 28;77(11):3173-3179. doi: 10.1093/jac/dkac299. PMID 36059138